CLINICAL TRIAL: NCT02695446
Title: Administration of Oral Extended Release Minocycline for Assessment of Skin and Plasma Concentrations of Minocycline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPX-01-C01
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral ER Minocycline - Up to 2mg/kg (Other): Oral extended release minocycline - up to 2mg/kg once a day for 30 days.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Oral extended release minocycline
  Other Names: MCN

SUMMARY:
The primary objective of this study is to evaluate the skin and plasma concentrations of minocycline in subjects undergoing treatment of acne vulgaris with oral extended release minocycline. Acne lesion counts and safety/tolerance of the treatment will also be evaluated.

DETAILED DESCRIPTION:
This will be an open label, non randomized, interventional pilot study evaluating the plasma and skin levels of minocycline in 10 subjects with moderate to severe acne vulgaris. Subjects with non inflammatory acne of nodular acne will not be enrolled. Subjects will be on an oral extended release minocycline regimen of up to 2mg/kg once a day for 4 weeks.

Steady state levels of minocycline in plasma and skin will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male and female subjects 14 to 40 years of age
* Moderate to severe inflammatory facial acne vulgaris (EGSA score of 3-5)
* Subjects not using oral or topical antibiotic products for at least 30 days prior to study entry and willing to refrain from use of oral and topical antibiotics for the duration of study participation
* Subjects not currently using and willing to refrain from use of other topical acne products for the duration of study participation

Exclusion Criteria:

* Mild, non-inflammatory or nodular acne vulgaris
* Have current or previous skin cancer
* Have a history of skin disease or presence of skin condition the PI believes would interfere with the study
* Females who report that they are pregnant, planning a pregnancy during the study period or breastfeeding
* Have conditions or factors that the PI believes may affect the response of the skin or the interpretation of the results
* Participation in any clinical study within the previous 30 days or plan concurrent participation in other studies

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lessin, MD, Principal Investigator — KGL, Inc.
Locations (1):
- KGL Skin Study Center, Broomall, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral ER Minocycline - Up to 2mg/kg
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral ER Minocycline - Up to 2mg/kg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 17 [14 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12
Plasma Minocycline (ng/ml) [Mean (Full Range); unit: ng/ml] | 0 [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Minocycline Level
Time Frame: Assessed at week 2 and week 4; reported at week 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Oral ER Minocycline - Up to 2mg/kg
Number analyzed (Participants) | 12
ng/ml | 421 (244)

2. Secondary Outcome: Skin/Dermal Levels of Minocycline
Time Frame: Measured at 2 weeks in half the subjects, 4 week biopsies not performed per early stopping rules
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Oral ER Minocycline - Up to 2mg/kg
Number analyzed (Participants) | 6
ng/ml | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Oral ER Minocycline - Up to 2mg/kg
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral ER Minocycline - Up to 2mg/kg (N=12)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No